CLINICAL TRIAL: NCT03839329
Title: Well-being in ACTion: Examining the Impact of Acceptance and Commitment Training in Community-Dwelling Older Adults
Brief Title: Group Acceptance and Commitment Training (ACT) With Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Roche, MA (Other)
Responsible Party: Sponsor-Investigator, Anne Roche, MA, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201902715
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Aging; Quality of Life
Keywords: Older Adult; Psychological Well-being; Acceptance and Commitment Therapy; Brief interventions; Psychological flexibility
MeSH Terms: conditions — Psychological Well-Being | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (stratified by sex) to either the ACT workshop group or to the assessment-only control group. Participants in the ACT group will complete two 90-minute group workshops (scheduled approximately one week apart) and will complete a baseline, 1-month, 3-month, and 6-month follow-up assessment. Participants in the time-matched assessment only-group will complete assessments at baseline, 1-month, 3-month, and 6-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Group Condition (Experimental): The ACT group condition will receive two 90-minute group Acceptance and Commitment Training (ACT) workshops (scheduled approximately one week apart) and will complete assessments.
  Interventions: Behavioral: Acceptance and Commitment Training
- Assessment-Only Condition (No Intervention): The Assessment-only condition will not receive any intervention and will only complete assessments.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Training — Acceptance and Commitment Therapy is an acceptance- and mindfulness-based psychotherapy that aims to foster psychological flexibility.
  Other Names: Acceptance and Commitment Therapy; ACT
  Arms: ACT Group Condition

SUMMARY:
The current study aims to explore the impact of a two-session group Acceptance and Commitment Therapy (ACT) intervention compared to an assessment-only control on psychological outcomes in healthy older adults. The proposed study has two main objectives.

1. Examine the impact the intervention on targeted ACT processes over time
2. Examine the impact of the intervention on aspects of eudaimonic well-being over time

DETAILED DESCRIPTION:
Older adults are a growing segment of our population, and this period of life presents a variety of physical, emotional, environmental, and cognitive changes, even for healthy individuals. The current study aims to explore the impact of a two-session group Acceptance and Commitment Therapy (ACT) intervention compared to an assessment-only control on psychological outcomes in healthy, community-dwelling older adults.

Participants will be randomly assigned (stratified by sex) to the ACT group condition or to an assessment-only control group. After randomization, those in the assessment-only control group will be asked to complete four assessments via mail (baseline, one-month, three-month, and six-month). The intervention group will participate in a brief group ACT intervention occurring over two sessions (90 minutes each, approximately one week apart). Intervention participants will also complete assessments at baseline and at one-month, three-months, and six-months post-intervention.

The specific aims and hypotheses of the current study are:

Specific Aim #1: To examine longitudinal between-group differences in targeted ACT processes including psychological flexibility (openness to experience, behavioral awareness, and valued action) and satisfaction with social roles and activities from baseline to follow-up. We hypothesize that there will be significant time by group interaction, such that psychological flexibility and satisfaction with social roles and activities will increase significantly more in the intervention group relative to the assessment-only control group.

Specific Aim #2: To examine longitudinal between-group differences in eudaimonic well-being (purpose in life and personal growth) from baseline to follow-up. We hypothesize that there will be significant time by group interactions, such that purpose in life and personal growth will increase significantly more in the intervention group relative to the assessment-only control group.

ELIGIBILITY:
Inclusion Criteria:

* healthy, community-dwelling older adult (age 65-99)

Exclusion Criteria:

* significant primary psychiatric disease
* medications that have the potential to affect cognitive functioning
* neurological events

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Differences in change over time between conditions on The Comprehensive Assessment of Acceptance and Commitment Therapy processes (CompACT) | baseline, 1-month, 3-month, and 6-month post-intervention follow-up
  The CompACT is a self-report measure of psychological flexibility. Total scores on the measure range from 0-138 with higher scores indicative of greater psychological flexibility.

SECONDARY OUTCOMES:
Differences in change over time between conditions on the Patient-Reported Outcomes Measurement Information System's (PROMIS) 8-item Satisfaction with Social Roles and Activities scale | baseline, 1-month, 3-month, and 6-month post-intervention follow-up
  The PROMIS 8-item Satisfaction with Social Roles and Activities scale is a self-report measure. Total scores on the measure are converted to T scores.
Differences in change over time between conditions on the Ryff's Scales of Psychological Well-Being 14-item Purpose in Life Scale | baseline, 1-month, 3-month, and 6-month post-intervention follow-up
  Ryff's Scales of Psychological Well-Being 14-item Purpose in Life Scale is a self-report measure. Total scores range from 14-84, with higher scores indicative of greater purpose in life.
Differences in change over time between conditions on the Ryff's Scales of Psychological Well-Being 14-item Personal Growth Scale | baseline, 1-month, 3-month, and 6-month post-intervention follow-up
  Ryff's Scales of Psychological Well-Being 14-item Personal Growth Scale is a self-report measure. Total scores range from 14-84, with higher scores indicative of greater personal growth.

CONTACTS AND LOCATIONS:
Overall Officials: Anne I Roche, MA, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No